CLINICAL TRIAL: NCT00782886
Title: Evaluation of Image-Guided Liver Surgical System for Resection of Liver Cancer
Status: Completed | Type: Observational
Sponsor: Pathfinder Therapeutics (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Medelis Inc., CRO
Other Study IDs: PTI-LC-2007-01; R44CA119502 (NIH)
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Liver Cancer
Keywords: Pathfinder; Liver; Resection; Surgery; To evaluate the effectiveness of image-guided liver surgery by measuring variables before, during and following surgery.; Completeness of resection and the accuracy of the resection, as determined by preoperative predicted RLV
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Image-guided surgery essentially describes the interactive use of medical images during a surgical procedure and is often referred to as a "global positioning" system (GPS) for surgery.

DETAILED DESCRIPTION:
In an automobile GPS, the current position of a vehicle is accurately localized or "registered" onto an electronic roadmap located on the dashboard. As the automobile moves, its position is updated on this roadmap. The driver can use the GPS as a guide to determine where the vehicle has been and where it is headed. This same concept is applied during image-guided surgery, as the current surgical position of instruments in the operating room is registered onto medical images of the patient acquired preoperatively. These images are used as a guide by the surgeon for more accurate localization of tumors and other surrounding anatomic structures. This clinical trial is designed to determine the effectiveness of using image-guided techniques for the treatment of liver tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained.
2. Patient must be 18 years or older.
3. Patients recruited are male or non-pregnant, non-lactating females. Liver resection or ablation could be harmful to an unborn child, and therefore is not recommended during pregnancy. All consented patients of childbearing potential will be advised to use adequate birth control (oral, implanted, or barrier methods), along with their sexual partners, while being considered for liver tumor resection or ablation and one month following surgery.
4. Negative serum or urine pregnancy test result at screening in women of childbearing potential (applies to patients without documented menopause or sterility).
5. Patients enrolled must be candidates for surgical liver resection of liver cancer (primary or metastatic) or benign liver lesions (hemangioma, Focal Nodular Hyperplasia, Adenoma). Liver cancer must be present on preoperative imaging study (CT and/or MRI), if applicable.
6. Patient must be scheduled for surgical treatment of the liver cancer requiring the removal of at least one (1) anatomic segment.

   -

Exclusion Criteria:

1. Any condition which, in the judgment of the clinical investigator or his designee, might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
2. Patients that have a mental condition rendering them unable to understand informed consent to the nature, scope, and possible consequences of this study.
3. Patients requiring surgical intervention that extends beyond the liver, with the exception that extension into some adjacent structures might be allowed unless the liver is not the primary focus of the surgery AND the potential blood loss from the other surgical sites may jeopardize the safety of the patient. There is no absolute rule as to what adjacent structures would be allowed, thus prior approval must be obtained from the Medical Monitor listed above for all extrahepatobiliary surgery.
4. Patients with hereditary hematologic/coagulation disorders unrelated to their liver disease.
5. Patients with cirrhosis of the liver classified as Child's B or C. (See Appendix A)
6. Use of aspirin within 7 days prior to surgery or antiplatelet agents (i.e., Plavix) within 10 days prior to surgery or nonsteroidal anti-inflammatory medications within 48 hours prior to surgery.
7. Patients with thrombocytopenia (platelet counts below 100,000 per ml, White Count 3.0, Hemoglobin 10 or greater).
8. Patients who are currently (within the last 30 days prior to surgery) participating in another clinical trial with any investigational drug or device.
9. Patients undergoing liver surgery as a result of trauma.
10. Patients undergoing liver surgery for the purpose of receiving a liver transplant.
11. Patients undergoing liver surgery in which there is a single minor wedge resection on the surface of the liver.
12. Patients with established renal insufficiency (defined as creatinine greater than 2.5 mg/dl), or a condition that requires hemodialysis.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving surgery for Liver disease.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The overall purpose of this NIH-funded study is to evaluate the effectiveness of image-guided liver surgery by measuring variables before, during and following surgery. | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: David Geller, M.D., Principal Investigator — UPMC Liver Cancer Center; William Jarnagin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Alan Hemming, M.D., Principal Investigator — University of Florida Department of Surgery
Locations (3):
- United States (3):
  - University of Florida Department of Surgery, Gainesville, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Pathfinder Therapeutics — http://www.2pti.com/
- See also: Medelis Inc. (CRO) — http://www.Medelis.com